CLINICAL TRIAL: NCT04098120
Title: Upper Gastrointestinal Endoscopic Findings In Chronic Kidney Disease And Haemodialyzed Patients In Assiut University Hospitals
Brief Title: Upper Endoscopy in CKD&ESRD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Abdelsalam Hasan, doctor, Assiut University
Other Study IDs: upper endoscopy in CKD&ESRD
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: CKD Stage(III,IV,V) and Haemodialyzed Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the study is To determine the necessity of upper gastrointestinal endoscopy in CKD(stage III---V) and haemodialyzed patients with upper GIT symptoms

DETAILED DESCRIPTION:
Chronic Kidney disease (CKD) is Kidney damage for ≥3 months, as defined by structural &or functional abnormalities of the kidney, with or without decreased GFR or GFR <60 mL/min/1.73m2 for ≥3 months, with or without kidney damage.

Stage Description GFR (ml/min/1.73 m2) Stage I Kidney damage >90 with normal or ↑ GFR Stage II Kidney damage with 60-89 mild ↓ in GFR Stage III Moderate ↓ in GFR 30-59 Stage IV Severe ↓ in GFR 15-29 Stage V Kidney failure < 15 < 15 (or dialysis) Or on dialysis

- CKD virtually affect the functions of all systems in our human body and associated with several deleterious effects on different systems which is due to multiple risk factors and associated with several abnormalities in the gastrointestinal tract involving all its segments, which include : Esophagitis: is present in more than a the third of the third of cases of uremic patients. It is due to increase of intra-abdominal pressure and reflux. The treatment of these patients is not different from that given to the general population with proton pump inhibitors, once the endoscopic study has been done.

Gastritis and peptic ulcer:as In patients with CKD and haemodialyzed patients, serum levels of gastrin are increased due to increased its secretion and decrease its excretion as it is eliminated by the kidney; additionally, cholecystokinin and secretin may be elevated. Noninvasive tests (H. pylori) have lower sensitivity in CKD so upper endscopy is needed.

In CKD and ESRD patients have more symptoms than general population.Specifically, gastrointestinal distress symptoms and peptic ulcers . The recurrence of peptic ulcer disease (PUD) after Helicobacter pylori eradication is higher in uremic patients than in non-uremic patients, and patients with ESRD have higher complication rates after ulcer development . Therefore, upper endoscopy should be performed in patients with these risk factors more often to prevent severe complications, such as gastrointestinal bleeding ( Haematemesis and melena). Angiodysplasia: affects the microcirculation of the mucosa and sub mucosa of the entire gastrointestinal tract. It is a frequent cause of bleeding in elderly patients, and its incidence is increased in patients on dialysis. Which diagnosed mainly by upper endoscopy as well as for the treatment with hemostasis techniques. The other option is angiography embolization, .

The manifestations of GIT in patients with chronic kidney disease and haemodialyzed patients varies from anorexia,nausea, vomiting they have aprevalance of around 60% )and GIT bleeding and viral hepatitis so it is across sectional study on 60 patients including CKD stage(III---V)and haemodialyzed patients.

* All patients will be subjected to :
* Full history and clinical examination . 2) Laboratory tests:

  1. CBC .
  2. liver function testes including PT,PC,INR
  3. blood urea and serum creatinine.
  4. serum calcium and phosphorus
  5. urine analysis. 3) abdominal ultrasonography 4) upper endoscopy

ELIGIBILITY:
Inclusion Criteria:

1.Patients with age varying from 20 to 60 years . 2.Patients diagnosed as CKD stage III - V and heamodialyzed patients . 3.presenting with upper GIT symptoms e.g anorexia,vomiting,melena…….etc

-

Exclusion Criteria:

1.Stage I and Stage II CKD patients. 2.Patients with uremic encephalopathy. 3.Patients undergone Renal transplant . 4.Patients with history of peptic disease. 5. patients on long time therapy with NSAIDs ,steroids. 6.patients with bleeding tendencies and coagulopathy. 7.Chronic alcoholic, Chronic Liver disease .

-

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: all CKD patients stage (III---V)and haemodialyzed patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Upper Gastrointestinal Endoscopic Findings In Chronic Kidney Disease And Haemodialyzed Patients | 2 years
  detect upper GIT complications as haematemesis and melena which threatening the life as ealy as possible